CLINICAL TRIAL: NCT04655300
Title: Evaluation of Age-related Skin Changes Using Clinical Probe Measurements and Imaging Modalities in Chinese Subjects
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-605-000
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Age-related Skin Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1
- Group 2
- Group 3
- Group 4
- Group 5
- Group 6

SUMMARY:
Evaluation of age-related skin changes using clinical probe measurements and imaging modalities in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects
* Subject agreeing to complete all study required procedures.
* Subject having given freely and expressly his/her informed consent.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or being in an exclusion period for a previous study.
* Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.
* Subject who underwent tissue augmentation with dermal fillers including HA, calcium hydroxylapatite, autologous fat, mesotherapy, or other cosmetic procedures (eg, face-lift, laser, photomodulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative procedures) in the face within 12 months before study entry or was planning to undergo any such treatment during the study.
* Subject who underwent treatment with botulinum toxins in the face or neck within 6 months of study entry or was planning to undergo such treatment during the study.
* Subject who ever received semi-permanent fillers or permanent facial implants (eg, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene) anywhere in the face or was planning to be implanted with any of these products at any time during the study.
* Subject with current cutaneous inflammatory or infectious processes (eg, acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion on the face that could interfere with measurements.
* Subject having changed, started or stopped any hormonal treatment or any treatment likely to have an impact on skin condition (over-the-counter or prescription, oral or topical, anti-wrinkle products on the face), within 30 days prior to enrollment or is planning to begin using such products during the study.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male Chinese subjects, between 20 and 79 years old, will be included in the study. Subjects will be divided in 6 age-categories: 20-29, 30-39, 40-49, 50-59, 60-69, 70-79 years (at least 10 subjects per decade and remainder of subjects distributed among the groups) in order to evaluate age-related skin changes.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Age-related changes in skin hydration on the cheeks, forehead, neck and around the mouth | 2 Months
  Skin hydration will be measured using tissue dielectric constant measurement. Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
Age-related changes in skin elasticity on the cheeks, forehead and neck | 2 Months
  Skin elasticity measurement using suction based device
Age-related changes in skin color on the cheeks and forehead | 2 Months
  Skin colorimetric measurement will be done with a Spectrophotometer
Age-related changes in skin thickness on the cheek | 2 Months
  Epidermal thickness will be measured with an optical coherence tomography instrument
Age-related changes in skin blood flow on the cheek | 2 Months
  Blood Flow (redness) will be measured with an optical coherence tomography instrument
Age-related changes in skin roughness on the cheek | 2 Months
  Skin surface roughness will be measured with an optical coherence tomography instrument
Age-related changes in skin OAC on the cheek | 2 Months
  Optical Attenuation Coefficient (OAC) will be measured with an optical coherence tomography instrument
Age-related changes in skin topography on the cheeks, forehead and around the mouth | 2 Months
  Skin topography imaged using a using a fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rq (Root Mean Square of the profile heights), RMax (Maximum Roughness Depth), Rv (Depth of the Largest Profile Valley), Rvm (Average depth of the Profile Valleys), Rz (average height of roughness) and Rt (maximum height of the roughness profile)
Age-related changes in gloss/shine, pores, skin color and texture on the cheek, forehead and around the mouth | 2 Months
  Skin gloss (Shine, pores, skin color and texture ) imaged using a camera-based system which uses various lighting/capture modalities to enhance the visualization of skin features
Clinical scoring of age-related changes in fine lines on the cheek | 2 Months
  The investigator will assess the participant's appearance of fine lines/wrinkles using a 5-point scale from (0=None to 4=Diffuse)
Clinical scoring of age-related changes in skin roughness on the cheek | 2 Months
  The investigator will assess the participant's appearance of skin roughness using a 5-point scale from (0=None to 4=Diffuse)

SECONDARY OUTCOMES:
To correlate the age-related skin hydration measurements on the cheeks, forehead, neck and around the mouth to clinical scoring of fine lines and skin smoothness. | 2 Months
  Skin hydration will be measured using tissue dielectric constant measurement. Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
To correlate the age-related skin elasticity measurements on the cheeks, forehead and neck to clinical scoring of fine lines and skin smoothness. | 2 Months
  Skin elasticity measurement using suction based device
To correlate the age-related skin color measurements on the cheeks and forehead to clinical scoring of fine lines and skin smoothness. | 2 Months
  Skin colorimetric measurement will be done with a Spectrophotometer
To correlate the age-related skin thickness measurements on the cheek to clinical scoring of fine lines and skin smoothness. | 2 Months
  Epidermal thickness will be measured with an optical coherence tomography instrument
To correlate the age-related skin blood flow measurements on the cheek to clinical scoring of fine lines and skin smoothness. | 2 Months
  Blood Flow (redness) will be measured with an optical coherence tomography instrument
To correlate the age-related skin roughness measurements on the cheek to clinical scoring of fine lines and skin smoothness. | 2 Months
  Skin surface roughness will be measured with an optical coherence tomography instrument
To correlate the age-related skin OAC measurements on the cheek to clinical scoring of fine lines and skin smoothness. | 2 Months
  Optical Attenuation Coefficient (OAC) will be measured with an optical coherence tomography instrument
To correlate the age-related skin topography measurements on the cheeks, forehead and around the mouth to clinical scoring of fine lines and skin smoothness. | 2 Months
  Skin topography imaged using a using a fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rq (Root Mean Square of the profile heights), RMax (Maximum Roughness Depth), Rv (Depth of the Largest Profile Valley), Rvm (Average depth of the Profile Valleys), Rz (average height of roughness) and Rt (maximum height of the roughness profile)
To correlate the age-related gloss/shine, pores, skin color and texture on the cheek, forehead and around the mouth to clinical scoring of fine lines and skin smoothness. | 2 Months
  Skin gloss (Shine, pores, skin color and texture ) imaged using a camera-based system which uses various lighting/capture modalities to enhance the visualization of skin features
To correlate the age-related fine lines on the cheek to clinical scoring of fine lines and skin smoothness. | 2 Months
  The investigator will assess the participant's appearance of fine lines/wrinkles using a 5-point scale from (0=None to 4=Diffuse)
To correlate the age-related skin roughness on the cheek to clinical scoring of fine lines and skin smoothness. | 2 Months
  The investigator will assess the participant's appearance of skin roughness using a 5-point scale from (0=None to 4=Diffuse)
Age-related changes and repeatability in the perioral area for hydration and topography. | 2 Months
  Skin hydration will be measured using tissue dielectric constant measurement. Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
  Skin topography imaged using a using a fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rq (Root Mean Square of the profile heights), RMax (Maximum Roughness Depth), Rv (Depth of the Largest Profile Valley), Rvm (Average depth of the Profile Valleys), Rz (average height of roughness) and Rt (maximum height of theroughness profile)
Age-related changes and repeatability in the neck for hydration and elasticity. | 2 Months
  Skin hydration will be measured using tissue dielectric constant measurement. Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
  Skin elasticity measurement using suction based device
Age related changes and repeatability in the forehead for hydration, color, elasticity, topography, skin gloss, color, texture, pores. | 2 Months
  Skin hydration will be measured using tissue dielectric constant measurement. Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
  Skin colorimetric measurement will be done with a Spectrophotometer. Skin elasticity measurement using suction based device. Skin topography imaged using a using a fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rq (Root Mean Square of the profile heights), RMax (Maximum Roughness Depth), Rv (Depth of the Largest Profile Valley), Rvm (Average depth of the Profile Valleys), Rz (average height of roughness) and Rt (maximum height of the roughness profile).
  Skin gloss (Shine, pores, skin color and texture ) imaged using a camera-based system which uses various lighting/capture modalities to enhance the visualization of skin features.

CONTACTS AND LOCATIONS:
Overall Officials: Min Liu, MD, Principal Investigator — Eurofins China
Locations (1):
- Eurofins China, Haizhu, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/search-results/?SearchTerm=NCT04655300&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&GenderDescriptions=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&hasResults=&isHighValue=&SortField=&SortOrder=